CLINICAL TRIAL: NCT01824277
Title: Diabetes Cardiac Surgery Initiative (DCI): A Community Based Pre-cardiac Surgery Diabetes Care Project
Brief Title: DCI: A Community Based Pre-cardiac Surgery Diabetes Care Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Rakesh C. Arora (Other)
Responsible Party: Sponsor-Investigator, Dr. Rakesh C. Arora, Medical Director, Intensive Care Cardiac Sciences, St. Boniface Hospital
Organization: St. Boniface Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GRT2012-53
Record Dates: First submitted 2013-03-31; First posted 2013-04-04 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (No Intervention): Group 1 - Standard Pre-operative Diabetes Care
- Group 2 (Experimental): Group 2 - Structured Pre-operative Diabetes Optimization
  Interventions: Other: Structured Pre-operative Diabetes Optimization

INTERVENTIONS:
Other: Structured Pre-operative Diabetes Optimization — Patients will receive structured pre-operative diabetes optimization while they wait for surgery. Patients will be referred to the Youville Diabetes Center where they will undergo preoperative optimization of their diabetes management. This will include in-depth diabetes education and instruction pertaining to lifestyle modification (blood glucose monitoring, nutrition, and physical activity) to improve glycemic control. Pharmacologic therapy will be reviewed by the Youville Diabetes Center certified diabetes nurse educators.
  Arms: Group 2

SUMMARY:
The Canadian Diabetes Association recommends optimizing glycemic control to achieve a glycated hemoglobin (A1C) of less than 7% in patients with diabetes. Despite these recommendations, approximately 25% of patients undergoing cardiac surgery have evidence of suboptimal glycemic control (A1C>7%). Recent research has demonstrated that such patients experience a higher rate of post-operative complications and significantly worse short-term and long-term post-operative survival. Therefore, it is recommended that attempts should be made to improve glycemic control while patients wait for their elective surgery. However, at present processes of care that facilitate pre-operative glycemic control optimization do not exist in Canada.

The objective of this project is to determine the feasibility and effectiveness of a comprehensive community-based pre-operative diabetes optimization program for patients awaiting elective cardiac surgery.

DETAILED DESCRIPTION:
This study is a randomized controlled trial and will investigate the feasibility and effectiveness of a pre-operative diabetes optimization program for patients with suboptimal glycemic control awaiting elective cardiac surgery. Consenting patients will be randomized to a Standard Pre-Operative Diabetes Care Group (Group 1) and a Structured Pre-Operative Diabetes Optimization Group (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand English
* Age > 18
* Able to provide informed consent
* A1C>7%
* Placed on the waiting list for elective cardiac surgery in Manitoba

Exclusion Criteria:

* Progressive cognitive deficit or disease.
* Age < 18
* Unable to provide informed consent
* A1C<7%
* Undergoing emergent cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in A1C over the study period. | Baseline to the patients' 3-months post-operative appointment

SECONDARY OUTCOMES:
Changes to the responses on the validated patient surveys | Baseline to the patients' 3-months post-operative appointment
  Surveys: Audit of Diabetes Quality of Life, Diabetes Treatment Satisfaction Questionnaire, and the SF-12 Health Related Quality of Life Questionnaire, Patient Health Questionnaire-9.
Changes in the patient perioperative outcomes | Baseline to the patients' 3-months post-operative appointment
  Surveys: Audit of Diabetes Quality of Life, Diabetes Treatment Satisfaction Questionnaire, and the SF-12 Health Related Quality of Life Questionnaire, Patient Health Questionnaire-9.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh C Arora, MD, Principal Investigator — University of Manitoba; Sora Ludwig, MD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Youville Diabetes Center, Winnipeg, Manitoba
  - I.H. AsperInstitute, St. Boniface General Hospital, Winnipeg, Manitoba